CLINICAL TRIAL: NCT01678729
Title: Does Pupil Size Matters in Refractive Surgery?
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0049-12-ZIV
Record Dates: First submitted 2012-08-30; First posted 2012-09-05 (Estimated); Last update posted 2012-09-05 (Estimated); Status verified 2012-08

CONDITIONS: Myopia
Keywords: refractive surgery; pupil; Pupil size
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
To determine the influence of pupil size in refractive surgery. If any influence exist.

ELIGIBILITY:
Inclusion Criteria:

- above 18 years suffers from myopia

Exclusion Criteria:

- suffer from keratoconus younger than 18 years old had previous eye surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: myopic patiens who did refractive surgery
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2009-01